CLINICAL TRIAL: NCT01222312
Title: Multicenter Randomized Phase II Study for the Therapy of Locally Advanced or Metastatic NSCLC (Stage IIIB/IV) With Cisplatin/Docetaxel or Oxaliplatin/Docetaxel
Brief Title: Study for Therapy of Locally Advanced or Metastatic Non Small Cell Lung Cancer (NSCLC) With Cisplatin / Docetaxel or Oxaliplatin / Docetaxel
Acronym: Taxelox
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S417
Record Dates: First submitted 2010-04-12; First posted 2010-10-18 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Non Small Cell Lung Cancer
Keywords: advanced NSCLC; oxaliplatin; cisplatin; docetaxel; locally advanced or metastatic non small cell lung cancer (stage IIIB-IV)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Oxaliplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A cisplatin (Active Comparator): Cisplatin 75 mg/m2, d1 Docetaxel 75 mg/m2, d1 every 3 weeks (d22) max. 6 cycles
  Interventions: Drug: Cisplatin; Drug: Docetaxel
- Arm B oxaliplatin (Experimental): Oxaliplatin 85 mg/m², d1 Docetaxel 50mg/m2, d1 every 2 weeks (d15) max. 8 cycles
  Interventions: Drug: Oxaliplatin; Drug: Docetaxel

INTERVENTIONS:
Drug: Cisplatin — 75 mg/m2, d1 every 3 weeks
  Arms: Arm A cisplatin
Drug: Oxaliplatin — 85 mg/m², d1 every 2 weeks
  Other Names: Eloxatin
  Arms: Arm B oxaliplatin
Drug: Docetaxel — 75 mg/m2, d1 every 3 weeks
  Other Names: Taxotere
  Arms: Arm A cisplatin
Drug: Docetaxel — 50mg/m2, d1 every 2 weeks
  Other Names: Taxotere
  Arms: Arm B oxaliplatin

SUMMARY:
The study compares two combinations of chemotherapy in patients with advanced or metastatic NSCLC: 50% of the patients are treated with cisplatin and docetaxel, the other 50% with oxaliplatin and docetaxel. cisplatin is today the standard therapy, but the toxicity profile is often not tolerable. Especially in elderly patients or patients with comorbidities, oxaliplatin based chemotherapy may have lower toxicities but comparable or even better response rates.

DETAILED DESCRIPTION:
Cispaltin based chemotherapies are standard for palliative first-line therapy in patients with advanced or metastatic NSCLC. Due to contraindications to cisplatin, this substance can not be used in a high number of patients. Especially in elderly patients, patients with comorbidities and patients with reduced general condition, cisplatin is a therapy which often induces intolerable toxicities. Thus, therapy often has to be interrupted or finished prematurely. Due to its favorable toxicity profile, oxaliplatin can be used also for the treatment of elderly patients and patients with comorbidities. Based on toxicity data from a phase II study of our group in patients with gastric cancer, the dosage for oxaliplatin/docetaxel was adopted for this actual study. In previous phase II trials, response rates of oxaliplatin based combination chemotherapies were comparable to those with cisplatin in patients with metastatic NSCLC.

In this study we will analyse, if a oxaliplatin based combination chemotherapy has a more tolerable toxicity profile and comparable or even better response rate in comparison to a cisplatin based chemotherapy. 44 patients in each arm will either be treated with a maximum of 6 cycles cisplatin/docetaxel or a maximum of 8 cycles oxaliplatin/docetaxel.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed NSCLC stage IIIB or IV.
* no previous chemotherapy in metastatic state
* male and female patients aged > 18 years
* ECOG ≤ 2
* Leukocytes > 3.000/µl
* Thrombocytes > 100.000/µl
* Serum creatinine ≤ 1.25x normal value, or Creatinine Clearance > 45 ml/min
* previous radiation < 25% bone marrow region allowed. Previous radiation of whole pelvis not allowed
* parallel radiation allowed, if target lesion outside of radiation field
* written informed consent
* life expectancy > 3 months

Exclusion Criteria:

* hypersensibility against Cisplatin, Oxaliplatin or Docetaxel
* Neoadjuvant or adjuvant chemotherapy within the last 6 months
* radiation within the last 28 days
* severe systemic comorbidities
* Cardiomyopathy or cardiac insufficiency stage II-IV according to NYHA
* malignant secondary disease, dated back < 5 years (exception: In-situ-carcinoma of the cervix uteri, adequately treated skin basal cell carcinoma)
* brain metastases
* severe non-surgical comorbidities or acute infection
* peripheral polyneuropathy > NCI grade II
* severe liver dysfunction AST/ALT>3,5xULN, AP>6xULN, Bilirubin>1,5xULN)
* participation in parallel trial
* pregnancy and lactation
* reduced hearing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2008-08; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
response rate | staging every 2 months

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | every two weeks
  comparison of adverse events (all grades, grade 3/4) in the Cisplatin vs Oxaliplatin arm
quality of life | every 8 weeks
progression free survival PFS | every 2 months
overall survival OS | 6 months follow-up
time to treatment failure TTF | every two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elke Jäger, Prof. Dr., Principal Investigator — Krankenhaus Nordwest
Locations (1):
- Krankenhaus Nordwest, Frankfurt am Main, Germany